CLINICAL TRIAL: NCT00911703
Title: Treatment Endpoints in Acute Decompensated Heart Failure
Brief Title: Determining When Patients Hospitalized With Acute Heart Failure Can Be Safely Sent Home (The DECIDE Study)
Acronym: DECIDE
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Abbott Point of Care (Industry); Inovise Medical (Industry)
Responsible Party: Principal Investigator, Sean Collins, Associate Proffesor of Emergency Medicine, Vanderbilt University
Other Study IDs: 659; K23HL085387-06 (NIH); K23HL085387-01A2 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2014-12

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute heart failure: Subjects with an ED diagnosis of acute decompensated heart failure .

SUMMARY:
The purpose of this study is to determine if certain findings (blood tests, symptom improvement, etc.) after acute heart failure treatment can identify a group of patients who are safe for early hospital discharge.

DETAILED DESCRIPTION:
A fundamental question faced by physicians treating acute decompensated heart failure (ADHF) is "When has treatment worked sufficiently for safe discharge, and who requires further treatment?" Patients with ADHF have a high incidence of morbidity and mortality. Current guidelines for emergency department (ED) and hospital disposition of patients with ADHF are based on limited empirical evidence. This creates clinical uncertainty regarding disposition leads to prolonged hospitalizations, higher costs and increased resource consumption. The specific aim of the study is to develop a prediction rule from readily available clinical data to help physicians identify ADHF patients eligible for safe and early discharge from the ED and hospital after treatment is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the modified Framingham criteria
* Have baseline data available within 1 hour of initial ED therapy
* Have previously documented systolic dysfunction (ejection fraction less than 50%) by echocardiogram
* Willing and able to give informed consent

The exclusion criteria are:

* Patients less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department who fulfill the modified Framingham criteria and are treated for acute heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 835 (Actual)
Dates: Start 2008-08; Primary Completion 2014-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Heart-failure related adverse events | Measured 5 days and 30 days after ED presentation

CONTACTS AND LOCATIONS:
Overall Officials: Sean P. Collins, MD, MSc, Principal Investigator — Vanderbilt University Emergency Medicine
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No